CLINICAL TRIAL: NCT05011409
Title: Prevalence of Depression and Anxiety Symptoms Among Newly Diagnosed Breast Cancer Patients in Almaty, Kazakhstan
Brief Title: Prevalence of Depression and Anxiety Among Breast Cancer Patients
Status: Completed | Type: Observational
Sponsor: Kazakh Medical University of Continuing Education (Other)
Collaborators: University of Malaya (Other)
Responsible Party: Sponsor
Other Study IDs: 06-2020
Record Dates: First submitted 2021-05-19; First posted 2021-08-18 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Depression; Anxiety; Breast Cancer
Keywords: depression; anxiety; breast cancer; prevalence; Beck Depression Inventory; Beck Anxiety Inventory
MeSH Terms: conditions — Depression; Anxiety Disorders; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly diagnosed breast cancer patients: Newly diagnosed breast cancer patients referred to Kazakh Institute of Oncology and Radiology or Almaty Oncology Center will be assessed on the prevalence of depression and anxiety symptoms.

SUMMARY:
Depression and anxiety in patients with breast cancer is serious comorbidity that affects the quality of life for patients, and their survival rates as they have poorer health outcomes. Furthermore, patients' high psychological burden is linked to higher healthcare costs. The investigation of the depression and anxiety symptoms prevalence among newly diagnosed breast cancer patients will help to navigate the health policy adjustment and psycho-social support system requirements. This study aims to investigate the prevalence of depression and anxiety symptoms among newly diagnosed breast cancer patients in Almaty, Kazakhstan, and associated risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Female adults with confirmed diagnosis of breast cancer within the 6 months study enrollment
* TNM stage I-IV
* Russian or Kazakh language proficiency
* Ability to provide informed consent

Exclusion Criteria:

* Current psychotic disorder, manic episode, serious neurological disorder, intellectual disability, or developmental disorder
* Current active suicidal ideation
* Referral to palliative care

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female breast cancer patients, not based on the self-representation of gender identity
Study Population: Study population will include breast cancer patients with confirmed diagnosis referred to the treatment to the Kazakh Institute of Oncology and Radiology and the Almaty Oncology Center
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2022-02-21 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of Depression Symptoms | within 6 months of diagnosis
  Prevalence of depression symptoms among newly diagnosed breast cancer patients according to the Beck Depression Inventory-II (BDI-II). The 21-item self-administered survey is scored on a scale of 0-3 in a list of four statements arranged in increasing severity about a particular symptom of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score for the Beck Depression Inventory-II (BDI-II). There is a four-point scale for each item ranging from 0 to 3. p. On two items (16 and 18) there are seven options to indicate either an increase or decrease of appetite and sleep. Cut-off score guidelines for the BDI-II are given with the recommendation that thresholds be adjusted based on the characteristics of the sample, and the purpose for use of the BDI-II. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Prevalence of Anxiety Symptoms | within 6 months of diagnosis
  Prevalence of anxiety symptoms among newly diagnosed breast cancer patients according to the Beck Anxiety Inventory. The Beck Anxiety Inventory (BAI) consists of 21 self-reported items (four-point scale ranging from 0 to 3. p.) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63).

CONTACTS AND LOCATIONS:
Overall Officials: Indira A Karibayeva, MPH, Principal Investigator — Kazakh Medical University of Continuing Education
Locations (2):
- Kazakhstan (2):
  - Almaty Oncology Center, Almaty
  - Kazakh Institute of Oncology and Radiology, Almaty

IPD SHARING:
Plan to Share IPD: Undecided
This plan is to be determined